CLINICAL TRIAL: NCT01058135
Title: A Randomized, Controlled, Double-blind Crossover Study to Assess the Effects of a Dietary Fiber Ingredient, at Two Doses, on Insulin Sensitivity
Brief Title: Effects of Hi-maize Resistant Starch on Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ingredion Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2010-09

CONDITIONS: Insulin Resistance
Keywords: insulin resistance; dietary fiber; resistant starch
MeSH Terms: conditions — Insulin Resistance | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Hi-maize starch (Low dose) — resistant starch
Other: Hi-maize starch (High-dose) — resistant starch
Other: Control (starch) — rapidly digestible starch

SUMMARY:
The purpose of this study is to determine the effects of a dietary fiber, resistant starch, on insulin sensitivity. Low insulin sensitivity is a risk factor for some diseases including type 2 diabetes and heart disease. This study will show if consuming resistant starch can help improve insulin sensitivity in overweight and obese people.

ELIGIBILITY:
Inclusion Criteria:

* Stable body weight
* No serious health conditions
* Waist circumference > or = to 89 cm (females) and 102 cm (males)

Exclusion Criteria:

* Diabetes
* other serious illnesses
* use of medications that affect outcomes
* BMI > or = 35.0 kg/m2

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | 4 weeks

SECONDARY OUTCOMES:
Inflammatory markers, glycemia, serum lipids | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Provident Clinical Research and Consulting, Inc, Glen Ellyn, Illinois, United States

REFERENCES:
- [Derived] Maki KC, Pelkman CL, Finocchiaro ET, Kelley KM, Lawless AL, Schild AL, Rains TM. Resistant starch from high-amylose maize increases insulin sensitivity in overweight and obese men. J Nutr. 2012 Apr;142(4):717-23. doi: 10.3945/jn.111.152975. Epub 2012 Feb 22. PMID 22357745
- See also: Related Info — http://www.resistantstarch.com